CLINICAL TRIAL: NCT03454555
Title: Integrated Health Services to Reduce Opioid Use While Managing Chronic Pain
Brief Title: Integrated Services for Pain: Interventions to Reduce Pain Effectively
Acronym: INSPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of North Carolina Health Care System (Unknown); Duke Health (Other); Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Lauren McCormack, Senior Vice President, RTI International
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCORI-OPD-1610-37006
Record Dates: First submitted 2018-02-27; First posted 2018-03-06 (Actual); Results first posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Chronic Pain
Keywords: Pragmatic Clinical Trial; Comparative Effectiveness Research; Analgesics, Opioid; Decision Making, Shared; Motivational Interviewing; Cognitive Therapy; Patient Reported Outcome Measures; Chronic Pain; Pain; Neurologic Manifestations
MeSH Terms: conditions — Chronic Pain; Pain; Neurologic Manifestations | interventions — Motivational Interviewing; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two intervention arms for the duration of the study. The study used real-time 1:1 ratio randomization to limit participant loss prior to treatment. Eligible patients were randomized using a stratified, permuted-block design, as this constrained randomization approach ensured balance between treatment groups within each of the 3 clinical institutions (the only stratification factor) at the completion of each block. Consequently, throughout the trial, the intervention arms were expected to have approximately equal sample sizes both within an institution and across the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shared Decision Making (SDM) (Active Comparator): Shared Decision Making (SDM) participants received guideline-concordant pharmacotherapy based on clinical guidelines for opioid therapy for chronic noncancer pain plus the SDM intervention during their opioid management visits.
  Interventions: Behavioral: Shared Decision Making
- Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) (Active Comparator): Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) participants received the guideline-concordant pharmacotherapy based on clinical guidelines for opioid therapy for chronic noncancer pain plus the MI+CBT-CP intervention.
  Interventions: Behavioral: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain

INTERVENTIONS:
Behavioral: Shared Decision Making — The Shared Decision Making (SDM) intervention is a patient-provider communication intervention to explore and compare treatment options, assess a patient's values and preferences, and reach a shared decision about chronic pain treatment. Participants in the SDM arm received their regular pain care visits with a designated SDM-trained clinician over a 12-month period. SDM intervention participants scheduled pain visits as often as needed for pain management (typically quarterly). SDM participants also received an electronic and physical packet of educational materials after randomization.
  Arms: Shared Decision Making (SDM)
Behavioral: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain — The Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) intervention is an empirically based behavioral pain management behavioral therapy intervention, including MI to enhance motivation for active participation in the CBT-CP, and the use of CBT-CP to enhance pain coping skills. MI + CBT-CP participants received one MI session plus up to eight weekly CBT-CP group sessions.
  Arms: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP)

SUMMARY:
Long-term pain -or pain that lasts for months or years-is one of the most common health problems in the United States. Clinicians often prescribe opioids which can help ease pain in the short term, but evidence does not support their effectiveness over the long term. For some people, long-term opioid use can lead to addiction and overdose. People need effective options and support to help maintain or improve their function and quality of life.

This study compared two programs for helping people living with long-term pain who have been prescribed opioids for 3 or more months. This study was done at primary care and pain care clinics at 3 health systems in the Southeastern United States.

The study team assigned people by chance to one of two study programs: (1) individual motivational interviewing plus group-based cognitive behavioral therapy (MI+CBT) or (2) patient-clinician shared decision making. In the MI+CBT program, the patient learned strategies to better cope with chronic pain. In the SDM program, the patient and clinician worked together through enhanced communication to make decisions that aligned with values and preferences of the patient.

The study team compared the two programs by looking at changes in opioid dosage, physical functioning, and pain interference over time. They collected information about prescribed opioid dosage from electronic health records and patients completed surveys at the start of the study and 6 and 12 months later.

The study team worked with an advisory group that included patients, advocates, clinicians, and pain experts. The advisory group met with the study team two to three times per year to provide input on the study.

DETAILED DESCRIPTION:
Objective:

To compare the effectiveness of individual motivational interviewing plus group-based cognitive behavioral therapy (MI+CBT) versus patient-clinician shared decision making (SDM) on change in daily dosage of prescribed opioids, physical functioning, and pain interference for individuals with chronic non-cancer pain (CNCP).

Rationale:

About 24% of Americans suffer from CNCP and clinicians often prescribe opioids to treat it. Once on chronic opioid therapy (COT), individuals often continue with this class of medication for years. Evidence for the effectiveness of COT to treat CNCP is limited, exposing individuals to known risks. Modified or novel pharmacological and nonpharmacological strategies are needed to improve pain management and promote informed decision making regarding possible opioid dose reduction.

Study Design and Approach:

This was a large-scale, pragmatic randomized controlled trial implementing pharmacotherapy guidelines and behavioral interventions in real-world settings. A key eligibility criterion was individuals who were prescribed ≥ 20 milligrams of morphine equivalents for more than three months.

Interventions:

Researchers examined the comparative effectiveness of MI+CBT versus SDM for who are on COT. Neither approach is directive, and both support patient choice. Although MI+CBT and SDM are both behavioral intervention strategies, they differ in content covered and training of those delivering the intervention (behavioral vs. medical). Participants in both study arms received guideline-concordant pharmacotherapy treatment, based on clinical guidelines for opioid therapy for CNCP.

Outcomes:

* Primary: The change from baseline in average daily prescribed opioid dosage, measured in milligrams of morphine equivalents, at 12 months, with secondary time points at 6 months and 18 months
* Secondary: The change from baseline to 6 and 12 months (primary timepoint) in the PROMIS Short Form v1.0 Pain Interference and PROMIS Short Form v1.0 Physical Function scales.

Timeline:

The project commenced in February 2018. Participant recruitment occurred from June 2019 to March 2022. Delivery of the intervention occurred on a rolling basis through March 2023.

Recruitment, Screening, Enrollment, and Randomization:

The study randomized 525 participants from primary care and pain clinics at three medical centers in North Carolina and Tennessee. The researchers identified individuals who were potentially eligible through electronic health records and invited them to participate. A Research Coordinator contacted individuals to complete screening, enrollment, and randomization.

Data Collection:

The researchers collected validated patient-reported outcomes through Web-based and phone-based surveys and leveraged existing harmonized electronic health record (EHR) data for clinical outcomes.

Data Analysis:

Outcomes were analyzed for all randomized participants in an intent-to-treat fashion, irrespective of the amount of intervention received. Because some individuals did not attend an intervention session, sensitivity analyses were based on a modified intent-to-treat population limited to participants receiving at least 1 intervention session and a per-protocol population limited to participants receiving at least four CBT or SDM sessions.

Changes from baseline were analyzed with a repeated measures linear model accounting for correlation of measurements over time, with effects for intervention arm, time interval as a categorical predictor, intervention-by-time interaction, and adjustment for baseline value and study site. Differential treatment effects for two preplanned subgroups based on sex and prior mental health diagnosis, as defined by IDC-10 codes recorded in the EHR, were assessed at 12 months via a subgroup-by-intervention interaction within the repeated measures model.

Qualitative research methods were used to obtain participant input on their experiences.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 85 years
* History of chronic non-cancer pain (CNCP)
* Receiving chronic opioid therapy for CNCP as evidenced by current or most recent prescription of an average daily prescribed dosage of 20 milligrams of morphine equivalents
* Receiving care at a participating clinic from a participating provider, as evidenced by at least 1 in-person visit within the past 12 months.

Exclusion Criteria:

* Not meeting the above inclusion criteria
* Opioid use is for pain directly related to an active cancer diagnosis
* Opioid use is for maintenance treatment of an opioid use disorder
* Suicide attempt within the past 3 years
* Active suicidal ideation
* Currently receiving Cognitive-Behavioral Therapy (CBT)
* Non-English speaking
* Other reason at the discretion of the investigator

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 543 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren McCormack, PhD, MSPH, Principal Investigator — RTI International
Locations (3):
- United States (3):
  - University of North Carolina Health Care System, Chapel Hill, North Carolina
  - Duke University Health System, Durham, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
RTI International plans to make available data from this study through the Patient-Centered Outcomes Data Repository (PCODR).
  The data package will include a de-identified copy of datasets containing all derived data used for all analysis and reporting.
Supporting Information: Study Protocol, SAP
Time Frame: Study data will be available for third-party requests when one of two conditions is met (whichever is met first):
  * The study funder, Patient-Centered Outcomes Research Institute (PCORI), makes the Final Research Report available on the PCORI website.
  * At the time of publication of the research project's primary results in a peer-reviewed journal.
  It is expected that data will be available until 7 years after RTI's contract with PCORI ends (2032).
Access Criteria: Third-party investigators seeking to access data will be required to complete and submit a data request form to PCODR. All requests for data will undergo review by an independent committee directed by PCODR staff. If the data request is approved, the data requestor's institution must enter into a Data Use Agreement (DUA). Approved data requestors will only have access to study data through a secure Virtual Data Enclave (VDE).
URL: http://www.pcori.org/sites/default/files/PCORI-Data-Management-and-Data-Sharing-Awardee-Guidance.pdf

REFERENCES:
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Chou R, Deyo R, Devine B, Hansen R, Sullivan S, Jarvik JG, Blazina I, Dana T, Bougatsos C, Turner J. The Effectiveness and Risks of Long-Term Opioid Treatment of Chronic Pain. Evid Rep Technol Assess (Full Rep). 2014 Sep;(218):1-219. doi: 10.23970/AHRQEPCERTA218. PMID 30313000
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Rose M, Bjorner JB, Gandek B, Bruce B, Fries JF, Ware JE Jr. The PROMIS Physical Function item bank was calibrated to a standardized metric and shown to improve measurement efficiency. J Clin Epidemiol. 2014 May;67(5):516-26. doi: 10.1016/j.jclinepi.2013.10.024. PMID 24698295
- [Background] Tan G, Jensen MP, Thornby JI, Shanti BF. Validation of the Brief Pain Inventory for chronic nonmalignant pain. J Pain. 2004 Mar;5(2):133-7. doi: 10.1016/j.jpain.2003.12.005. PMID 15042521
- [Background] Amtmann D, Cook KF, Jensen MP, Chen WH, Choi S, Revicki D, Cella D, Rothrock N, Keefe F, Callahan L, Lai JS. Development of a PROMIS item bank to measure pain interference. Pain. 2010 Jul;150(1):173-182. doi: 10.1016/j.pain.2010.04.025. PMID 20554116
- [Background] Bann CM, McCormack LA, Berkman ND, Squiers LB. The Health Literacy Skills Instrument: a 10-item short form. J Health Commun. 2012;17 Suppl 3(Suppl 3):191-202. doi: 10.1080/10810730.2012.718042. PMID 23030570
- [Background] Boonstra AM, Schiphorst Preuper HR, Balk GA, Stewart RE. Cut-off points for mild, moderate, and severe pain on the visual analogue scale for pain in patients with chronic musculoskeletal pain. Pain. 2014 Dec;155(12):2545-2550. doi: 10.1016/j.pain.2014.09.014. Epub 2014 Sep 17. PMID 25239073
- [Background] Edlund MJ, Thomas SM, Wagner LK, Thompson JE, Wu LT, Dolor RJ, Chelminski PR, Ives TJ, Archer KR, Dewey CM, Sullivan MD, McCormack LA; INSPIRE Study Team. Design of a Multicenter Randomized Controlled Trial comparing the effectiveness of shared decision making versus motivational interviewing plus cognitive behavioral therapy for voluntary opioid tapering: The INSPIRE study protocol. Contemp Clin Trials. 2024 Feb;137:107410. doi: 10.1016/j.cct.2023.107410. Epub 2023 Dec 12. PMID 38092285
- [Background] Martin BC, Fan MY, Edlund MJ, Devries A, Braden JB, Sullivan MD. Long-term chronic opioid therapy discontinuation rates from the TROUP study. J Gen Intern Med. 2011 Dec;26(12):1450-7. doi: 10.1007/s11606-011-1771-0. Epub 2011 Jul 13. PMID 21751058
- [Background] Monticone M, Ambrosini E, Cedraschi C, Rocca B, Fiorentini R, Restelli M, Gianola S, Ferrante S, Zanoli G, Moja L. Cognitive-behavioral Treatment for Subacute and Chronic Neck Pain: A Cochrane Review. Spine (Phila Pa 1976). 2015 Oct 1;40(19):1495-504. doi: 10.1097/BRS.0000000000001052. PMID 26192729
- [Background] Rose M, Bjorner JB, Becker J, Fries JF, Ware JE. Evaluation of a preliminary physical function item bank supported the expected advantages of the Patient-Reported Outcomes Measurement Information System (PROMIS). J Clin Epidemiol. 2008 Jan;61(1):17-33. doi: 10.1016/j.jclinepi.2006.06.025. PMID 18083459
- [Background] Vanderlip ER, Sullivan MD, Edlund MJ, Martin BC, Fortney J, Austen M, Williams JS, Hudson T. National study of discontinuation of long-term opioid therapy among veterans. Pain. 2014 Dec;155(12):2673-2679. doi: 10.1016/j.pain.2014.09.034. Epub 2014 Sep 30. PMID 25277462
- [Result] McCormack LA, Edlund MJ, Thomas SM, Wu LT, Chelminski PR, Archer KR, Wagner LK, Hirsch S, Thompson JE, Dolor RJ, Ives TJ, Dewey CM, Chang S; INSPIRE Study Team. Effectiveness of motivational interviewing plus cognitive behavioral therapy vs shared decision making for voluntary opioid tapering in patients with chronic pain: the INSPIRE randomized pragmatic trial. Pain Med. 2025 Aug 1;26(8):477-489. doi: 10.1093/pm/pnaf049. PMID 40338272
- [Result] Chang SH, Hirsch SC, Thomas SM, Edlund MJ, Dolor RJ, Ives TJ, Dewey CM, Gulur P, Chelminski PR, Archer KR, Wu LT, Curtis J, Goldstein AO, McCormack LA; INSPIRE Study Team. Complexities and approaches for deriving longitudinal daily morphine milligram equivalents using electronic health record prescription data. JAMIA Open. 2025 Jun 16;8(3):ooaf053. doi: 10.1093/jamiaopen/ooaf053. eCollection 2025 Jun. PMID 40524838
- See also: Study description on research team's organizational website — https://www.rti.org/impact/inspire-trial-managing-long-term-pain
- See also: Institute of Medicine (US) Committee on Advancing Pain Research, Care, and Education. Relieving Pain in America: A Blueprint for Transforming Prevention, Care, Education, and Research. Washington (DC): National Academies Press (US); 2011. — https://nap.nationalacademies.org/catalog/13172/relieving-pain-in-america-a-blueprint-for-transforming-prevention-care
- See also: Study description on funder's website — https://www.pcori.org/research-results/2017/comparing-two-ways-help-patients-manage-long-term-non-cancer-pain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 3 academic health systems between June 26, 2019 and March 31, 2022.
Pre-assignment Details: Of 543 consented participants, 525 were randomized to treatment. Of those not randomized, 7 were lost to follow-up, 6 were determined ineligible after consent, 1 withdrew consent, 2 were withdrawn by an investigator, and 2 were not randomized for reasons unknown.
Groups:
- Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP): Motivational Interviewing (MI) and Cognitive Behavioral Therapy for Chronic Pain (CBT-CP) [MI+CBT-CP] participants received the guideline-concordant pharmacotherapy based on clinical guidelines for opioid therapy for chronic noncancer pain plus the MI+CBT-CP intervention. MI+CBT-CP participants received one MI session plus up to eight weekly CBT-CP group sessions.
- Shared Decision Making (SDM): Shared Decision Making (SDM) participants received guideline-concordant pharmacotherapy based on clinical guidelines for opioid therapy for chronic noncancer pain plus the SDM intervention during their opioid management visits. Participants in the SDM arm received their regular pain care visits with a designated SDM-trained clinician over a 12-month period. SDM intervention participants scheduled pain visits as often as needed for pain management (typically quarterly). SDM participants also received an electronic and physical packet of educational materials after randomization.
Period: Overall Study
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM)
Started | 263 | 262
Completed | 189 | 228
Not Completed | 74 | 34
Not completed — Death | 6 | 6
Not completed — Lost to Follow-up | 31 | 12
Not completed — Physician Decision | 2 | 6
Not completed — Withdrawal by Subject | 34 | 5
Not completed — Ineligible | 1 | 5

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) population
Groups:
- Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP): Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) participants received the guideline-concordant pharmacotherapy based on clinical guidelines for opioid therapy for chronic noncancer pain plus the MI+CBT-CP intervention. MI + CBT-CP participants received one MI session plus up to eight weekly CBT-CP group sessions.
- Total: Total of all reporting groups
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM) | Total
Number analyzed (Participants) | 263 | 262 | 525
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age was unknown or not reported for 8 participants.
  years
    number analyzed (Participants) | 259 | 258 | 517
    (all) | 57.4 (11.3) | 58.6 (11.6) | 58.0 (11.5)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex at Birth: Female | 167 | 163 | 330
  Sex at Birth: Male | 93 | 99 | 192
  Sex at Birth: Missing | 3 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 252 | 254 | 506
  Unknown or Not Reported | 6 | 2 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 67 | 57 | 124
  Race: White | 170 | 182 | 352
  Race: Other | 11 | 12 | 23
  Race: Multiracial | 11 | 9 | 20
  Race: Missing | 4 | 2 | 6
Study Site [Count of Participants; unit: Participants]
  University of North Carolina at Chapel Hill (UNC) | 87 | 86 | 173
  Duke University | 91 | 90 | 181
  Vanderbilt University Medical Center (VUMC) | 85 | 86 | 171
Education [Count of Participants; unit: Participants]
  High school degree (or General Education Diploma [GED]) or less | 72 | 86 | 158
  Some college or a 2-year degree | 100 | 97 | 197
  Bachelor's degree or more | 89 | 79 | 168
  Missing | 2 | 0 | 2
Health Literacy Level [Count of Participants; unit: Participants] — The Health Literacy Skills Instrument was used to assess participant health literacy in terms of print literacy (reading and writing), numeracy skills, oral literacy skills (listening), and information seeking (navigation of Internet and facilities). The version used in the study had 5 questions.
  Health literacy level was classified into 3 categories: High Health Literacy (all 5 questions correct), Average Health Literacy (3 or 4 questions correct), and Low Health Literacy (0 to 2 questions correct). Missing responses were counted as incorrect.
  Participants
    High | 97 | 89 | 186
    Average | 114 | 114 | 228
    Low | 50 | 59 | 109
    Missing | 2 | 0 | 2
Employment Status [Count of Participants; unit: Participants]
  Working part- or full-time | 55 | 42 | 97
  Not employed, retired | 57 | 64 | 121
  Not employed for health reasons or disabled | 143 | 140 | 283
  Other (looking for work, in school, homemaker) | 6 | 16 | 22
  Missing | 2 | 0 | 2
Body Mass Index [Count of Participants; unit: Participants]
  Obese (BMI >=30) | 158 | 142 | 300
  Not Obese (BMI < 30) | 105 | 120 | 225
Average Daily Opioid Dose (in Morphine Milligram Equivalents [MME]) [Median (Inter-Quartile Range); unit: Morphine Milligram Equivalents] — Average daily opioid dose was derived from electronic health records. Dose is reported in morphine milligram equivalents (MME), a standardized measure that accounts for differences in opioid prescription strength, quantity, and potency relative to morphine. Baseline average daily opioid dose was calculated as the prescribed daily MME averaged over the 90 days prior to randomization. Higher MME values indicate greater opioid dosage prescribed. Population: Eleven participants did not have an opioid prescription during the baseline period (defined as 3 months before enrollment): 5 had an opioid prescribed at an outside clinic and later transferred to the study clinic, 4 received an opioid just before the baseline period, and 2 received a type of opioid (e.g., injectable) that was not included in the study.
  Morphine Milligram Equivalents
    number analyzed (Participants) | 257 | 257 | 514
    (all) | 59 [26 to 108] | 50 [29 to 90] | 53 [28 to 99]
Average Daily Opioid Dose Categories [Count of Participants; unit: Participants]
  None | 6 | 5 | 11
  Very Low (<20 MME) | 26 | 24 | 50
  Low (20 - <50 MME) | 93 | 104 | 197
  Moderate (50 - <90 MME) | 52 | 64 | 116
  High (90+ MME) | 86 | 65 | 151
Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference T-Score [Mean (Standard Deviation); unit: units on a scale (T-Score)] — The PROMIS Pain Interference 8-item scale is a validated, self-reported instrument assessing pain interference over the past 7 days. Pain interference is a measure of the extent to which pain interferes with patient physical, mental, and social activities. Responses were scored using the PROMIS scoring system to generate a standardized T-score, allowing comparison to the general population (mean = 50, standard deviation = 10). Higher T-scores indicate higher pain interference and worse health.
  units on a scale (T-Score) | 65.8 (5.9) | 65.9 (6.0) | 65.8 (5.9)
PROMIS Physical Functioning T-Score [Mean (Standard Deviation); unit: units on a scale (T-Score)] — The PROMIS Physical Functioning measure is a validated, self-reported instrument assessing physical functioning over the past 7 days. Physical functioning measures one's upper extremities (dexterity), lower extremities (walking and mobility), central regions (back and neck), and instrumental activities of daily living. Responses were scored using the PROMIS scoring system to generate a standardized T-score, allowing comparison to the general population (mean = 50, SD = 10). Higher T-scores indicate higher physical functioning and better health.
  units on a scale (T-Score) | 34.4 (6.0) | 35.1 (6.3) | 34.7 (6.2)
Brief Pain Index (BPI) Pain Severity [Count of Participants; unit: Participants] — The BPI Pain Severity scale is a validated, self-reported measure assessing pain severity at its worst and least in the past 7 days, on average, and right now. Possible scores on each item range from 0 (no pain) to 10 (pain as bad as you can imagine). Higher scores indicate higher pain severity and worse health. The scores were averaged to generate a composite score from 0 to 10. BPI pain severity categories are defined as Mild (0 to 3.5), Moderate (3.5 to 7.4), and Severe (7.5 to 10).
  Participants
    Missing | 2 | 0 | 2
    Mild | 3 | 10 | 13
    Moderate | 189 | 176 | 365
    Severe | 69 | 76 | 145
Presence of 1+ Comorbid Mental Health Diagnoses [Count of Participants; unit: Participants] — Presence of any of the following mental health disorder diagnoses in the participant's electronic health record: adjustment disorder, anxiety, attention-deficit/hyperactivity disorder, dementia, developmental disorder, childhood disorders, impulse control disorder, mood disorder, personality disorder, schizophrenia or other psychotic disorder, suicidal ideation, and other miscellaneous mental health disorders.
  Participants
    Yes | 119 | 108 | 227
    No | 144 | 154 | 298
Charlson Comorbidity Index (CCI) categories based on diagnosis codes [Count of Participants; unit: Participants] — Presence of any of the following conditions in the participant's electronic health record: myocardial infarction, congestive heart failure, peripheral vascular disease, cerebrovascular disease, dementia, chronic pulmonary disease, rheumatic disease, peptic ulcer disease, mild liver disease, diabetes without complications, diabetes with complications, paraplegia and hemiplegia, renal disease, cancer, moderate or severe liver disease, metastatic carcinoma, or AIDS/HIV. These conditions make up the Charlson Comorbidity Index, a measure of overall health status and mortality risk.
  Participants
    None | 128 | 135 | 263
    1 or more CGI Index Categories | 135 | 127 | 262
Presence of Substance Use Disorder Diagnosis Code [Count of Participants; unit: Participants] — Presence of any substance use disorder diagnoses in the participant's electronic health record.
  Participants
    Yes | 66 | 69 | 135
    No | 197 | 193 | 390

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Daily Opioid Dose in Morphine Milligram Equivalents (MME) at Month 12
Description: The primary outcome was derived from electronic health records. Total morphine equivalents for each prescription was calculated by multiplying the quantity of each prescription by the strength of the prescription (milligrams of opioid per unit dispensed). The quantity-strength product was then multiplied by conversion factors to estimate the milligrams of morphine equivalent to the opioids dispensed in the prescription. The total average dose in morphine equivalents per day supplied was calculated by summing the morphine equivalents for each prescription filled during a given period and dividing by the number of days supplied. Opioid dose was calculated as the prescribed milligrams of daily morphine equivalent dose averaged over the 90 days prior to randomization and averaged over 90 days for the time period of 12 months post-randomization. Change in daily opioid dose was computed as the difference between the dose calculated during that period and the dose from the baseline period.
Time Frame: Month 12 (PRIMARY TIMEPOINT)
Population: Intent-to-treat population; those missing EHR prescription data at a certain timepoint did not contribute data for that timepoint in the mixed repeated measures model.
Measure: Least Squares Mean (95% Confidence Interval); unit: Morphine Milligram Equivalents (MME)
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM)
Number analyzed (Participants) | 220 | 223
Morphine Milligram Equivalents (MME) | -11.6 [-19.1 to -4.1] | -6.0 [-14.0 to 2.0]
Statistical Analysis 1: Comparison: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) vs Shared Decision Making (SDM); Test type: Superiority; p = 0.31, Mixed Models Analysis; Mean Difference (Final Values) = -5.6, 95% CI 2-sided [-16.6 to 5.3]

2. Primary Outcome: Change From Baseline in Average Daily Opioid Dose in Morphine Milligram Equivalents (MME) at Month 3
Description: The primary outcome was derived from electronic health records. Total morphine equivalents for each prescription was calculated by multiplying the quantity of each prescription by the strength of the prescription (milligrams of opioid per unit dispensed). The quantity-strength product was then multiplied by conversion factors to estimate the milligrams of morphine equivalent to the opioids dispensed in the prescription. The total average dose in morphine equivalents per day supplied was calculated by summing the morphine equivalents for each prescription filled during a given period and dividing by the number of days supplied. Opioid dose was calculated as the prescribed milligrams of daily morphine equivalent dose averaged over the 90 days prior to randomization and averaged over 90 days for the time period of 3 months post-randomization. Change in daily opioid dose was computed as the difference between the dose calculated during that period and the dose from the baseline period.
Time Frame: Month 3
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Morphine Milligram Equivalents (MME)
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM)
Number analyzed (Participants) | 254 | 253
Morphine Milligram Equivalents (MME) | 0.0 [-7.2 to 7.1] | -0.3 [-8.0 to 7.4]
Statistical Analysis 1: Comparison: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) vs Shared Decision Making (SDM); Test type: Superiority; p = 0.963, Mixed Models Analysis; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-10.3 to 10.7]

3. Primary Outcome: Change From Baseline in Average Daily Opioid Dose in in Morphine Milligram Equivalents (MME) at Month 6
Description: The primary outcome was derived from electronic health records. Total morphine equivalents for each prescription was calculated by multiplying the quantity of each prescription by the strength of the prescription (milligrams of opioid per unit dispensed). The quantity-strength product was then multiplied by conversion factors to estimate the milligrams of morphine equivalent to the opioids dispensed in the prescription. The total average dose in morphine equivalents per day supplied was calculated by summing the morphine equivalents for each prescription filled during a given period and dividing by the number of days supplied. Opioid dose was calculated as the prescribed milligrams of daily morphine equivalent dose averaged over the 90 days prior to randomization and averaged over 90 days for the time period of 6 months post-randomization. Change in daily opioid dose was computed as the difference between the dose calculated during that period and the dose from the baseline period.
Time Frame: Month 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Morphine Milligram Equivalents (MME)
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM)
Number analyzed (Participants) | 238 | 247
Morphine Milligram Equivalents (MME) | -5.9 [-13.2 to 1.4] | 0.3 [-7.4 to 8.1]
Statistical Analysis 1: Comparison: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) vs Shared Decision Making (SDM); Test type: Superiority; p = 0.253, Mixed Models Analysis; Mean Difference (Final Values) = -6.2, 95% CI 2-sided [-16.8 to 4.4]

4. Primary Outcome: Change From Baseline in Average Daily Opioid Dose in Morphine Milligram Equivalents (MME) at Month 9
Description: The primary outcome was derived from electronic health records. Total morphine equivalents for each prescription was calculated by multiplying the quantity of each prescription by the strength of the prescription (milligrams of opioid per unit dispensed). The quantity-strength product was then multiplied by conversion factors to estimate the milligrams of morphine equivalent to the opioids dispensed in the prescription. The total average dose in morphine equivalents per day supplied was calculated by summing the morphine equivalents for each prescription filled during a given period and dividing by the number of days supplied. Opioid dose was calculated as the prescribed milligrams of daily morphine equivalent dose averaged over the 90 days prior to randomization and averaged over 90 days for the time period of 9 months post-randomization. Change in daily opioid dose was computed as the difference between the dose calculated during that period and the dose from the baseline period.
Time Frame: Month 9
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Morphine Milligram Equivalents (MME)
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM)
Number analyzed (Participants) | 228 | 236
Morphine Milligram Equivalents (MME) | -6.6 [-14.0 to 0.8] | -7.3 [-15.1 to 0.6]
Statistical Analysis 1: Comparison: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) vs Shared Decision Making (SDM); Test type: Superiority; p = 0.90, Mixed Models Analysis; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-10.1 to 11.5]

5. Primary Outcome: Change From Baseline in Average Daily Opioid Dose in Morphine Milligram Equivalents (MME) at Month 15
Description: The primary outcome was derived from electronic health records. Total morphine equivalents for each prescription was calculated by multiplying the quantity of each prescription by the strength of the prescription (milligrams of opioid per unit dispensed). The quantity-strength product was then multiplied by conversion factors to estimate the milligrams of morphine equivalent to the opioids dispensed in the prescription. The total average dose in morphine equivalents per day supplied was calculated by summing the morphine equivalents for each prescription filled during a given period and dividing by the number of days supplied. Opioid dose was calculated as the prescribed milligrams of daily morphine equivalent dose averaged over the 90 days prior to randomization and averaged over 90 days for the time period of 15 months post-randomization. Change in daily opioid dose was computed as the difference between the dose calculated during that period and the dose from the baseline period.
Time Frame: Month 15
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Morphine Milligram Equivalents (MME)
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM)
Number analyzed (Participants) | 206 | 216
Morphine Milligram Equivalents (MME) | -9.4 [-17.1 to -1.7] | -6.8 [-14.9 to 1.2]
Statistical Analysis 1: Comparison: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) vs Shared Decision Making (SDM); Test type: Superiority; p = 0.65, Mixed Models Analysis; Mean Difference (Final Values) = -2.6, 95% CI 2-sided [-13.7 to 8.6]

6. Primary Outcome: Change From Baseline in Average Daily Opioid Dose in Morphine Milligram Equivalents (MME) at Month 18
Description: The primary outcome was derived from electronic health records. Total morphine equivalents for each prescription was calculated by multiplying the quantity of each prescription by the strength of the prescription (milligrams of opioid per unit dispensed). The quantity-strength product was then multiplied by conversion factors to estimate the milligrams of morphine equivalent to the opioids dispensed in the prescription. The total average dose in morphine equivalents per day supplied was calculated by summing the morphine equivalents for each prescription filled during a given period and dividing by the number of days supplied. Opioid dose was calculated as the prescribed milligrams of daily morphine equivalent dose averaged over the 90 days prior to randomization and averaged over 90 days for the time period of 18 months post-randomization. Change in daily opioid dose was computed as the difference between the dose calculated during that period and the dose from the baseline period.
Time Frame: Month 18
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Morphine Milligram Equivalents (MME)
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM)
Number analyzed (Participants) | 197 | 197
Morphine Milligram Equivalents (MME) | -3.1 [-10.9 to 4.8] | -12.5 [-20.7 to -4.4]
Statistical Analysis 1: Comparison: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) vs Shared Decision Making (SDM); Test type: Superiority; p = 0.102, Mixed Models Analysis; Mean Difference (Final Values) = 9.4, 95% CI 2-sided [-1.9 to 20.8]

7. Primary Outcome: Change From Baseline of at Least 10 Morphine Milligram Equivalents (MME) at Month 12
Description: Dichotomous variable indicating a decrease of 10 MME or more from baseline to 12 months (1=yes and 0 =no). Modeled the probability of having a 10 or more MME decrease from baseline.
Time Frame: Month 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Estimated proportion
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM)
Number analyzed (Participants) | 220 | 223
Estimated proportion | 0.29 [0.20 to 0.38] | 0.30 [0.22 to 0.40]
Statistical Analysis 1: Comparison: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) vs Shared Decision Making (SDM); Test type: Superiority; p = 0.83, Mixed Models Analysis; Used a logistic mixed model for repeated measures; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.50 to 1.75]

8. Primary Outcome: Change From Baseline of at Least 10 Morphine Milligram Equivalents (MME) at Month 3
Description: as for outcome 7
Time Frame: Month 3
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Estimated proportion
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM)
Number analyzed (Participants) | 254 | 253
Estimated proportion | 0.13 [0.09 to 0.20] | 0.16 [0.11 to 0.23]
Statistical Analysis 1: Comparison: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) vs Shared Decision Making (SDM); Test type: Superiority; p = 0.47, Mixed Models Analysis; Used a logistic mixed model for repeated measures; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.42 to 1.50]

9. Primary Outcome: Change From Baseline of at Least 10 Morphine Milligram Equivalents (MME) at Month 6
Description: as for outcome 7
Time Frame: Month 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Estimated proportion
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM)
Number analyzed (Participants) | 238 | 247
Estimated proportion | 0.21 [0.14 to 0.29] | 0.21 [0.14 to 0.29]
Statistical Analysis 1: Comparison: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) vs Shared Decision Making (SDM); Test type: Superiority; p = 0.96, Mixed Models Analysis; Used a logistic mixed model for repeated measures; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.54 to 1.90]

10. Primary Outcome: Change From Baseline of at Least 10 Morphine Milligram Equivalents (MME) at Month 9
Description: as for outcome 7
Time Frame: Month 9
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Estimated proportion
Groups:
- Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP): MI+CBT-CP participants will receive the guideline-concordant pharmacotherapy based on clinical guidelines for opioid therapy for chronic noncancer pain plus the MI+CBT-CP intervention.
  Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain: The Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) intervention is an empirically based behavioral pain management behavioral therapy intervention, including MI to enhance motivation for active participation in the CBT-CP, and the use of CBT-CP to enhance pain coping skills. One individual MI session will focus on patient engagement and enhancing a patient's own intrinsic motivation for CBT-CP participation. MI will also be woven into the group CBT-CP sessions. We will deliver 8 sessions of CBT-CP, as is standard in a group setting, in-person or virtually.
- Shared Decision Making (SDM): SDM participants will receive guideline-concordant pharmacotherapy based on clinical guidelines for opioid therapy for chronic noncancer pain plus the SDM intervention during their opioid management visits.
  Shared Decision Making: The Shared Decision Making (SDM) intervention is a patient-provider communication intervention to explore and compare treatment options, assess a patient's values and preferences, and reach a shared decision about chronic pain treatment. The intervention will have both clinician and patient educational components. The content of the clinician component will be based on the Agency for Healthcare Research and Quality's "SHARE: Seek, Help, Assess, Reach, Evaluate" Approach, which is a 5-step process for shared decision making that includes exploring and comparing the benefits, harms, and risks of each option through meaningful dialogue about what matters most to the patient. Participants randomized to Arm 1 will have their study visits and opioid use managed by an SDM-trained clinician at their practice.
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM)
Number analyzed (Participants) | 228 | 236
Estimated proportion | 0.22 [0.15 to 0.31] | 0.28 [0.20 to 0.38]
Statistical Analysis 1: Comparison: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) vs Shared Decision Making (SDM); Test type: Superiority; p = 0.28, Mixed Models Analysis; Used a logistic mixed model for repeated measures; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.38 to 1.33]

11. Primary Outcome: Change From Baseline of at Least 10 Morphine Milligram Equivalents (MME) at Month 15
Description: as for outcome 7
Time Frame: Month 15
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Estimated proportion
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM)
Number analyzed (Participants) | 206 | 216
Estimated proportion | 0.30 [0.21 to 0.41] | 0.32 [0.23 to 0.42]
Statistical Analysis 1: Comparison: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) vs Shared Decision Making (SDM); Test type: Superiority; p = 0.75, Mixed Models Analysis; Used a logistic mixed model for repeated measures; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.47 to 1.71]

12. Primary Outcome: Change From Baseline of at Least 10 Morphine Milligram Equivalents (MME) at Month 18
Description: as for outcome 7
Time Frame: Month 18
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Estimated proportion
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM)
Number analyzed (Participants) | 197 | 197
Estimated proportion | 0.26 [0.18 to 0.37] | 0.35 [0.25 to 0.46]
Statistical Analysis 1: Comparison: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) vs Shared Decision Making (SDM); Test type: Superiority; p = 0.25, Mixed Models Analysis; Used a logistic mixed model for repeated measures; Odds Ratio (OR) = 0.68, 95% CI 2-sided [0.35 to 1.31]

13. Secondary Outcome: Change From Baseline in Pain Interference on the 8-item Patient-Reported Outcomes Measurement Information System - Pain Interference (PROMIS-PI) at Month 6
Description: The Patient-Reported Outcomes Measurement Information System - Pain Interference (PROMIS-PI) is a validated, self-reported instrument assessing pain interference over the past 7 days. Pain interference is a measure of the extent to which pain interferes with patient physical, mental, and social activities. Possible scores on each item range in value from 1 (not at all) to 5 (very much). Higher T-scores indicate higher pain interference and worse health. Change = Month 6 Score - Baseline Score.
Time Frame: Month 6
Population: Intent-to-treat population among those that completed a 6-month survey. 1 participant in the SDM arm did not complete the entire 6-month survey, but did complete the PROMIS Pain Interference section of the survey and was included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale (T-score)
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM)
Number analyzed (Participants) | 142 | 159
units on a scale (T-score) | 0.5 [-0.4 to 1.4] | 0.3 [-0.4 to 1.0]
Statistical Analysis 1: Comparison: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) vs Shared Decision Making (SDM); Test type: Superiority; p = 0.70, Mixed Models Analysis; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.9 to 1.4]

14. Secondary Outcome: Change From Baseline in Pain Interference on the 8-item Patient-Reported Outcomes Measurement Information System - Pain Interference (PROMIS-PI) at Month 12
Description: The Patient-Reported Outcomes Measurement Information System - Pain Interference (PROMIS-PI) is a validated, self-reported instrument assessing pain interference over the past 7 days. Pain interference is a measure of the extent to which pain interferes with patient physical, mental, and social activities. Possible scores on each item range in value from 1 (not at all) to 5 (very much). Higher T-scores indicate higher pain interference and worse health. Change = Month 12 Score - Baseline Score.
Time Frame: Month 12
Population: Intent-to-treat population among those that completed a 12-month survey. 1 participant in the CBT arm and 5 in the SDM arm did not complete the entire 12-month survey, but did complete the PROMIS Pain Interference section of the survey and were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale (T-score)
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM)
Number analyzed (Participants) | 130 | 157
units on a scale (T-score) | 0.1 [-0.8 to 1.0] | 0.0 [-0.7 to 0.7]
Statistical Analysis 1: Comparison: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) vs Shared Decision Making (SDM); Test type: Superiority; p = 0.92, Mixed Models Analysis; Median Difference (Final Values) = 0.1, 95% CI 2-sided [-1.1 to 1.2]

15. Secondary Outcome: Change From Baseline in Physical Functioning on the 8-item Patient-Reported Outcomes Measurement Information System - Physical Functioning (PROMIS-PF) at Month 6
Description: The Patient-Reported Outcomes Measurement Information System - Physical Functioning (PROMIS-PF) is a validated, self-reported instrument assessing physical functioning over the past 7 days. Physical functioning measures one's upper extremities (dexterity), lower extremities (walking and mobility), central regions (back and neck), and instrumental activities of daily living.
  Possible scores on each item range in value from 1 (without any difficulty) to 5 (unable to do). Higher T-scores indicate higher physical functioning and better health. Change = Month 6 Score - Baseline Score.
Time Frame: Month 6
Population: Intent-to-treat population among those that completed a 6-month survey.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale (T-score)
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM)
Number analyzed (Participants) | 142 | 158
units on a scale (T-score) | -0.4 [-1.1 to 0.3] | -0.6 [-1.3 to 0.1]
Statistical Analysis 1: Comparison: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) vs Shared Decision Making (SDM); Test type: Superiority; p = 0.64, Mixed Models Analysis; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.7 to 1.2]

16. Secondary Outcome: Change From Baseline in Physical Functioning on the 8-item Patient-Reported Outcomes Measurement Information System - Physical Functioning (PROMIS-PF) at Month 12
Description: The Patient-Reported Outcomes Measurement Information System - Physical Functioning (PROMIS-PF) is a validated, self-reported instrument assessing physical functioning over the past 7 days. Physical functioning measures one's upper extremities (dexterity), lower extremities (walking and mobility), central regions (back and neck), and instrumental activities of daily living.
  Possible scores on each item range in value from 1 (without any difficulty) to 5 (unable to do). Higher T-scores indicate higher physical functioning and better health. Change = Month 12 Score - Baseline Score.
Time Frame: Month 12
Population: Intent-to-treat population among those that completed a 12-month survey. 1 participant in the CBT arm and 5 in the SDM arm did not complete the entire 12-month survey, but did complete the PROMIS Physical Functioning section of the survey and were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale (T-score)
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM)
Number analyzed (Participants) | 130 | 157
units on a scale (T-score) | -0.3 [-1.0 to 0.4] | -0.5 [-1.1 to 0.2]
Statistical Analysis 1: Comparison: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) vs Shared Decision Making (SDM); Test type: Superiority; p = 0.75, Mixed Models Analysis; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.8 to 1.1]

17. Other Pre Specified Outcome: Change From Baseline in Pain Intensity on the 3-item Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity at Month 6
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS)-Pain Intensity is a validated, self-reported instrument assessing pain intensity over the past 7 days. Possible scores on each item range in value from 1 (no pain) to 5 (very severe). Higher T-scores indicate higher pain intensity and worse health. Change = Month 6 Score - Baseline Score.
Time Frame: Month 6
Population: Intent-to-treat population among those that completed a 6-month survey. 1 participant in the SDM arm did not complete the entire 6-month survey, but did complete the PROMIS Pain Intensity section of the survey and was included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale (T-score)
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM)
Number analyzed (Participants) | 141 | 159
units on a scale (T-score) | -0.8 [-1.6 to 0.1] | -1.0 [-1.8 to -0.2]
Statistical Analysis 1: Comparison: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) vs Shared Decision Making (SDM); Test type: Superiority; p = 0.69, Mixed Models Analysis; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.9 to 1.4]

18. Other Pre Specified Outcome: Change From Baseline in Pain Intensity on the 3-item Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity at Month 12
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity is a validated, self-reported instrument assessing pain intensity over the past 7 days. Possible scores on each item range in value from 1 (no pain) to 5 (very severe). Higher T-scores indicate higher pain intensity and worse health. Change = Month 12 Score - Baseline Score.
Time Frame: Month 12
Population: Intent-to-treat population among those that completed a 12-month survey. 1 participant in the CBT arm and 3 in the SDM arm did not complete the entire 12-month survey, but did complete the PROMIS Pain Intensity section of the survey and were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale (T-score)
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM)
Number analyzed (Participants) | 130 | 155
units on a scale (T-score) | -0.9 [-1.8 to 0.0] | -1.5 [-2.3 to -0.7]
Statistical Analysis 1: Comparison: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) vs Shared Decision Making (SDM); Test type: Superiority; p = 0.33, Mixed Models Analysis; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-0.6 to 1.8]

19. Other Pre Specified Outcome: Change From Baseline in Anxiety on the 4-item Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress - Anxiety at Month 6
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress-Anxiety is a validated, self-reported instrument assessing anxiety over the past 7 days. Anxiety measures self-reported fear, anxiety, hyperarousal, and somatic symptoms related to arousal. Anxiety is best differentiated by symptoms that reflect autonomic arousal and experience of threat. Possible scores on each item range in value from 1 (never) to 5 (always). Higher T-scores indicate higher anxiety and worse health. Change = Month 6 Score - Baseline Score.
Time Frame: Month 6
Population: Intent-to-treat population among those that completed a 6-month survey. 1 participant in the SDM arm did not complete the entire 6-month survey, but did complete the PROMIS Anxiety section of the survey and was included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale (T-score)
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM)
Number analyzed (Participants) | 142 | 159
units on a scale (T-score) | 1.7 [0.6 to 2.8] | 1.8 [0.7 to 3.0]
Statistical Analysis 1: Comparison: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) vs Shared Decision Making (SDM); Test type: Superiority; p = 0.86, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-1.8 to 1.5]

20. Other Pre Specified Outcome: Change From Baseline in Anxiety on the 4-item Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress - Anxiety at Month 12
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress-Anxiety is a validated, self-reported instrument assessing anxiety over the past 7 days. Anxiety measures self-reported fear, anxiety, hyperarousal, and somatic symptoms related to arousal. Anxiety is best differentiated by symptoms that reflect autonomic arousal and experience of threat. Possible scores on each item range in value from 1 (never) to 5 (always). Higher T-scores indicate higher anxiety and worse health. Change = Month 12 Score - Baseline Score.
Time Frame: Month 12
Population: Intent-to-treat population among those that completed a 12-month survey. 3 participants in the SDM arm did not complete the entire 12-month survey, but did complete the PROMIS Anxiety section of the survey and were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale (T-score)
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM)
Number analyzed (Participants) | 128 | 155
units on a scale (T-score) | 1.9 [0.8 to 3.1] | 1.7 [0.5 to 2.9]
Statistical Analysis 1: Comparison: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) vs Shared Decision Making (SDM); Test type: Superiority; p = 0.76, Mixed Models Analysis; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-1.4 to 1.9]

21. Other Pre Specified Outcome: Change From Baseline in Depression on the 4-item Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress-Depression at Month 6
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS)-Emotional Distress-Depression is a validated, self-reported instrument assessing depression over the past 7 days. Depression measures self-reported negative mood, views of self, social cognition, and decreased positive affect and engagement. Possible scores on each item range in value from 1 (never) to 5 (always). Higher T-scores indicate higher depression and worse health. Change = Month 6 Score - Baseline Score.
Time Frame: Month 6
Population: Intent-to-treat population among those that completed a 6-month survey.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale (T-score)
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM)
Number analyzed (Participants) | 142 | 158
units on a scale (T-score) | 1.3 [0.2 to 2.3] | 1.7 [0.6 to 2.8]
Statistical Analysis 1: Comparison: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) vs Shared Decision Making (SDM); Test type: Superiority; p = 0.55, Mixed Models Analysis; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-2.0 to 1.1]

22. Other Pre Specified Outcome: Change From Baseline in Depression on the 4-item Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress-Depression at Month 12
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS)-Emotional Distress-Depression is a validated, self-reported instrument assessing depression over the past 7 days. Depression measures self-reported negative mood, views of self, social cognition, and decreased positive affect and engagement. Possible scores on each item range in value from 1 (never) to 5 (always). Higher T-scores indicate higher depression and worse health. Change = Month 12 Score - Baseline Score.
Time Frame: Month 12
Population: Intent-to-treat population among those that completed a 12-month survey. 3 participants in the SDM arm did not complete the entire 12-month survey, but did complete the PROMIS Depression section of the survey and were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale (T-score)
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM)
Number analyzed (Participants) | 129 | 155
units on a scale (T-score) | 1.5 [0.4 to 2.6] | 2.0 [0.9 to 3.1]
Statistical Analysis 1: Comparison: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) vs Shared Decision Making (SDM); Test type: Superiority; p = 0.52, Mixed Models Analysis; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-2.1 to 1.1]

23. Other Pre Specified Outcome: Change From Baseline in Pain Severity on the 4-item Brief Pain Inventory (BPI) Pain Severity at Month 6
Description: The Brief Pain Inventory (BPI) Pain Severity is a validated, self-reported instrument assessing pain severity at its worst and least in the past 7 days, on average, and right now. Possible scores on each item range from 0 (no pain) to 10 (pain as bad as you can imagine). Higher scores indicate higher pain severity and worse health. Change = Month 6 Score - Baseline Score.
Time Frame: Month 6
Population: Intent-to-treat population among those that completed a 6-month survey.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM)
Number analyzed (Participants) | 142 | 158
units on a scale | -0.1 [-0.3 to 0.1] | -0.2 [-0.4 to 0.0]
Statistical Analysis 1: Comparison: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) vs Shared Decision Making (SDM); Test type: Superiority; p = 0.37, Mixed Models Analysis; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.2 to 0.4]

24. Other Pre Specified Outcome: Change From Baseline in Pain Severity on the 4-item Brief Pain Inventory (BPI) Pain Severity at Month 12
Description: The Brief Pain Inventory (BPI) Pain Severity is a validated, self-reported instrument assessing pain severity at its worst and least in the past 7 days, on average, and right now. Possible scores on each item range from 0 (no pain) to 10 (pain as bad as you can imagine). Higher scores indicate higher pain severity and worse health. Change = Month 12 Score - Baseline Score.
Time Frame: Month 12
Population: Intent-to-treat population among those that completed a 12-month survey. 3 participants in the SDM arm did not complete the entire 12-month survey, but did complete the BPI Pain Severity section of the survey and were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM)
Number analyzed (Participants) | 129 | 155
units on a scale | -0.2 [-0.4 to 0.0] | -0.2 [-0.4 to 0.0]
Statistical Analysis 1: Comparison: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) vs Shared Decision Making (SDM); Test type: Superiority; p = 0.91, Mixed Models Analysis; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.3 to 0.3]

25. Other Pre Specified Outcome: Change From Baseline in Pain Interference on the 7-item Brief Pain Inventory (BPI) Pain Interference at Month 6
Description: The Brief Pain Inventory (BPI) Pain Interference is a validated, self-reported instrument assessing pain interference over the past 7 days in 7 categories: general activity, walking, work, mood, enjoyment of life, relation with others, and sleep. Possible scores on each item range from 0 (does not interfere) to 10 (completely interferes). Higher scores indicate higher pain interference and worse health. Change = Month 6 Score - Baseline Score.
Time Frame: Month 6
Population: Intent-to-treat population among those that completed a 6-month survey.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM)
Number analyzed (Participants) | 142 | 158
units on a scale | 0.0 [-0.3 to 0.3] | -0.2 [-0.5 to 0.0]
Statistical Analysis 1: Comparison: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) vs Shared Decision Making (SDM); Test type: Superiority; p = 0.33, Mixed Models Analysis; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.2 to 0.6]

26. Other Pre Specified Outcome: Change From Baseline in Pain Interference on the 7-item Brief Pain Inventory (BPI) Pain Interference at Month 12
Description: The Brief Pain Inventory (BPI) Pain Interference is a validated, self-reported instrument assessing pain interference over the past 7 days in 7 categories: general activity, walking, work, mood, enjoyment of life, relation with others, and sleep. Possible scores on each item range from 0 (does not interfere) to 10 (completely interferes). Higher scores indicate higher pain interference and worse health. Change = Month 12 Score - Baseline Score.
Time Frame: Month 12
Population: Intent-to-treat population among those that completed a 12-month survey. 3 participants in the SDM arm did not complete the entire 12-month survey, but did complete the BPI Pain Interference section of the survey and were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM)
Number analyzed (Participants) | 129 | 155
units on a scale | 0.1 [-0.2 to 0.4] | -0.1 [-0.2 to 0.2]
Statistical Analysis 1: Comparison: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) vs Shared Decision Making (SDM); Test type: Superiority; p = 0.46, Mixed Models Analysis; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.3 to 0.6]

27. Other Pre Specified Outcome: Discontinuation of Opioid Medications at Month 12
Description: Discontinuation of opioid medications at Month 12 was assessed with a self-reported item newly developed for this study and electronic health record (EHR) data. Discontinuation was defined as a response of "No" to a question on the Month 12 participant survey that asked: "Are you currently taking an opioid medicine now? Commonly prescribed opioids include hydrocodone, oxycodone, codeine, morphine, and fentanyl" AND no opioid prescriptions in the EHR within 15 days prior to Month 12 through Month 18.
Time Frame: Month 12
Population: Intent-to-treat population and those that completed the 12-month survey; 2 participants in the SDM arm did not complete the entire 12-month survey but did complete the self-report use of opioid medication section and were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM)
Number analyzed (Participants) | 129 | 154
Participants
  Taking an opioid prescription at 12 months | 119 | 145
  Discontinued opioid prescription at 12 months | 10 | 9
Statistical Analysis 1: Comparison: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) vs Shared Decision Making (SDM); Test type: Superiority; p = 0.52, Chi-squared; Risk Difference (RD) = -0.02, 95% CI 2-sided [-0.08 to 0.04]

28. Other Pre Specified Outcome: Intent to Taper at Month 6
Description: Intent to Taper was assessed with a self-reported item, newly developed for this study, that assessed intent to reduce the amount of opioids taken: "Please say how much you agree with this statement: 'Reducing the amount of opioid medicines I take is a goal of mine.'" Possible response options included Strongly Agree, Agree, Uncertain, Disagree, and Strongly Disagree. Responses of Strongly Agree or Agree were categorized as an intent to taper, and responses of Uncertain, Disagree, Strongly Disagree, or Don't Know were categorized as no intent to taper.
Time Frame: Month 6
Population: Intent-to-treat population among those that completed this specific question on the 6-month survey. If participant reported not currently taking an opioid at the 6-month survey, this question was skipped.
Measure: Least Squares Mean (95% Confidence Interval); unit: Estimated proportion
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM)
Number analyzed (Participants) | 123 | 135
Estimated proportion | 0.66 [0.56 to 0.74] | 0.56 [0.47 to 0.65]
Statistical Analysis 1: Comparison: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) vs Shared Decision Making (SDM); Test type: Superiority; p = 0.17, Mixed Models Analysis; Used a generalized logistic model for repeated measurements; modeled the outcome of intention to taper; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.85 to 2.59]

29. Other Pre Specified Outcome: Intent to Taper at Month 12
Description: as for outcome 28
Time Frame: Month 12
Population: Intent-to-treat population among those that completed this specific question on the 12-month survey. If participant reported not currently taking an opioid at the 12-month survey, this question was skipped.
Measure: Least Squares Mean (95% Confidence Interval); unit: Estimated proportion
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM)
Number analyzed (Participants) | 108 | 130
Estimated proportion | 0.62 [0.52 to 0.72] | 0.57 [0.47 to 0.66]
Statistical Analysis 1: Comparison: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) vs Shared Decision Making (SDM); Test type: Superiority; p = 0.41, Mixed Models Analysis; Used a generalized logistic model for repeated measurements; modeled the outcome of intention to taper; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.71 to 2.31]

30. Other Pre Specified Outcome: Relative Opioid Use Self-report at Month 6
Description: Opioid use relative to baseline was assessed with a self-reported item, newly developed for this study: "Since you started taking part in this study, would you say that your overall use of opioids has increased, stayed about the same, or decreased? In thinking about your "overall use" we ask you consider how often you take the opioid medicine, the different types of opioid medicines, and their amounts." Possible response options included: My overall use of opioids has increased; My overall use of opioids has stayed about the same; and My overall use of opioids has decreased.
Time Frame: Month 6
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM)
Number analyzed (Participants) | 122 | 135
Participants
  Opioid Use Increased since Study Start | 13 | 13
  Opioid Use Stayed About the Same since Study Start | 83 | 89
  Opioid Use Decreased since Study Start | 26 | 33
Statistical Analysis 1: Comparison: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) vs Shared Decision Making (SDM); Test type: Superiority; p = 0.79, Chi-squared

31. Other Pre Specified Outcome: Relative Opioid Use Self-report at Month 12
Description: as for outcome 30
Time Frame: Month 12
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) | Shared Decision Making (SDM)
Number analyzed (Participants) | 108 | 130
Participants
  Opioid Use has Increased since Study Start | 8 | 10
  Opioid Use has Stayed about the Same since Study Start | 71 | 92
  Opioid Use has Decreased since Study Start | 29 | 28
Statistical Analysis 1: Comparison: Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) vs Shared Decision Making (SDM); Test type: Superiority; p = 0.67, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse Events were reported from baseline through the 12-month intervention phase of the study.
Description: Study adverse event (AE) reporting was limited to 4 types of events: suicide ideation (active suicidal ideation or attempted suicide), opioid withdrawal, opioid overdose, and death. AEs were collected by study coordinators, self-reported on surveys at 6 and 12 months, and by electronic health record International Classification of Diseases, Tenth Revision (ICD-10) codes.
  Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Shared Decision Making (SDM) | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP)
All-Cause Mortality (participants affected / at risk) | 6/262 | 6/263
Serious Adverse Events (participants affected / at risk) | 21/262 | 17/263
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Shared Decision Making (SDM) (N=262) | Motivational Interviewing and Cognitive Behavioral Therapy for Chronic Pain (MI+CBT-CP) (N=263)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 2 (2)
Death (General disorders) | 6 (6) | 6 (6)
Opioid Overdose (Psychiatric disorders) | 4 (4) | 2 (2)
Opioid Withdrawal (Psychiatric disorders) | 9 (12) | 8 (9)

LIMITATIONS AND CAVEATS:
Academic medical centers as study sites may limit applicability to other settings. Patients mostly on low or medium opioid doses. INSPIRE was conducted during the peak of coronavirus disease 2019 (COVID-19). Technological barriers could have hindered participation. Clinicians and patients may have been reluctant to taper opioids during telehealth visits. Pandemic-related hardships may have affected self-reported quality of life measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/55/NCT03454555/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/55/NCT03454555/SAP_001.pdf